CLINICAL TRIAL: NCT02515019
Title: Bispectral Index Guided Titration of Sevoflurane in On-pump Cardiac Surgery Reduces Plasma Sevoflurane Concentration and Vasopressor Requirements
Brief Title: Bispectral Index Guided Sevoflurane Titration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. med. Rainer Nitzschke, Dr. Rainer Nitzschke, Universitätsklinikum Hamburg-Eppendorf
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sevo_2_2014
Record Dates: First submitted 2015-07-28; First posted 2015-08-04 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Intraoperative Hypotension
Keywords: Anaesthetics inhalation; Bispectral index; Cardiopulmonary bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Sevo1.8% (No Intervention): Anaesthesia was maintained with a constant inspired concentration of sevoflurane 1.8% (Sevorane; Abbvie, Wiesbaden, Germany) administered via the ventilator. From the beginning of CPB, a constant flow of sevoflurane 1.8% was administered with the oxygenator fresh-gas supply, using a common anaesthetic vaporiser (Draeger Vapor Version 2000; Draeger, Luebeck, Germany). Following successful weaning from CPB, sevoflurane was again administered at an inspired concentration of 1.8% using the ventilator.
- Bispectral index Monitoring (Experimental): The sevoflurane concentration via the ventilator and the oxygenator fresh gas supply was titrated to maintain a target BIS value between 40 and 60 (BIS-Monitor, Covidien, Boulder, Colorado, USA). However, the concentration of sevoflurane in the oxygenator fresh gas supply was not reduced below 0.3%.
  Interventions: Device: Bispectral index Monitoring

INTERVENTIONS:
Device: Bispectral index Monitoring — In group SevoBIS, the sevoflurane concentration was titrated to maintain a target BIS value between 40 and 60.
  Other Names: BIS-Monitor, Covidien, Boulder, Colorado, USA
  Arms: Bispectral index Monitoring

SUMMARY:
Electroencephalographic-based monitoring systems such as the bispectral index (BIS) may reduce anaesthetic overdose rates. The investigators hypothesised that goal-directed sevoflurane administration (guided by BIS monitoring) could reduce the sevoflurane plasma concentration (SPC) and intraoperative vasopressor doses during on-pump cardiac surgery in a prospective, controlled, sequential two-arm clinical study.

DETAILED DESCRIPTION:
Electroencephalographic (EEG)-based monitoring systems, for example the bispectral index [(BIS); BIS monitor, Covidien, Boulder, Colorado, USA], were designed to prevent anaesthesia underdosage with the risk of awareness and to reduce the time to awakening after terminating general anaesthesia. However, little is known about the consequences of anaesthetic overdose. The investigators assume that high doses of anaesthetics result in cardiocirculatory depression and the necessity for high-dose vasopressor therapy, followed by microcirculation disorder and organ dysfunction.

The investigators hypothesised that in on-pump cardiac-surgery, goaldirected administration of sevoflurane guided by BIS monitoring reduces excessive sevoflurane plasma concentration (SPC) and the need for an intraoperative vasopressor. To test this hypothesis, the current study compared BIS-guided sevoflurane administration with the constant delivery of an inspired sevoflurane concentration of 1.8% during on-pump cardiac surgery and analysed its effect on the SPC and the required intraoperative dosage of norepinephrine.

The study population was divided into two patient groups: Thirty-three on-pump cardiac surgery patients enrolled in the study were allocated to a conventionally treated control group, with the constant administration of an inspired concentration of sevoflurane 1.8% (group Sevo1.8%). Thirty-four patients were sequentially allocated to an interventional group with BIS-guided administration of sevoflurane (group SevoBIS).

Vasoactive drugs were administered according to the following protocol in both groups. If the mean arterial blood pressure decreased below 50 mmHg, a continuous infusion of norepinephrine was given to maintain a perfusion pressure between 50 and 60 mmHg during cardiopulmonary bypass. If the mean arterial pressure increased above 75 mmHg, nitroglycerine was used in boluses of 0.1 mg until arterial pressure returned to a mean of less than 75 mmHg. If mean arterial pressure persisted above 75 mmHg after a cumulative administration of nitroglycerine 1.0 mg, urapidil was administered in boluses of 0.1 mg/kg until the perfusion pressure decreased below 75 mmHg.

At the end of the surgical procedure, all patients were transferred to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective on-pump cardiac surgery and an American Society of Anesthesiologists' (ASA) physical status of 3 to 4

Exclusion Criteria:

* A contraindication to the administration of volatile anaesthetics, an active infection with a temperature more than 38°C and any history of neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Cumulative intraoperative administration of norepinephrine | During operation

SECONDARY OUTCOMES:
Sevoflurane concentration in the oxygenator freshgas supply during cardiopulmonary bypass | During operation
Postoperative blood lactate concentration | Upon arrival in the intensive care unit (ICU)
Duration of postoperative mechanical ventilation | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
ICU length of stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Incidence of acute kidney injury | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Sevoflurane Plasma Concentration during CPB | During operation

CONTACTS AND LOCATIONS:
Overall Officials: Christian Zoellner, Professor, Study Chair — Department of Anesthesiology; Center of Anesthesiology and Intensive Care Medicine, Hamburg Eppendorf University Medical Center
Locations (1):
- Department of Anesthesiology; Center of Anesthesiology and Intensive Care Medicine, Hamburg Eppendorf University Medical Center, Hamburg, Germany

REFERENCES:
- See also: Publication of study results - Bispectral index guided titration of sevoflurane in on-pump cardiac surgery reduces plasma sevoflurane concentration and vasopressor requirements: A prospective, controlled, sequential two-arm clinical study — https://journals.lww.com/ejanaesthesiology/fulltext/2014/09000/Bispectral_index_guided_titration_of_sevoflurane.7.aspx#pdf-link